CLINICAL TRIAL: NCT03637894
Title: Immunity Modification of Full Term Infants According to the Type of Feeding and Mode of Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Heinz Italia SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FERT15
Record Dates: First submitted 2018-01-11; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-01

CONDITIONS: Innate Immunity; Newborns; Nutrition; Microbiota
Keywords: Newborns; Fermented milk; Innate immunity

STUDY DESIGN:
Intervention Model Description: RCT double blind study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Infants born by CS-fed fermented formula (Active Comparator): Feeding infants with fermented formula milk. Infants born by cesarean section were fed either with fermented formula milk or with standard formula during the first 3 months of life
  Interventions: Dietary Supplement: Feeding infants with fermented formula milk
- Infants born by CS-fed standard formula (Placebo Comparator): Feeding infants with standard formula milk. Infants born by cesarean section were fed either with fermented formula milk or with standard formula during the first 3 months of life
  Interventions: Other: Feeding infants with standard formula milk
- Infants born by CS-breastfed (Other): Infants born by cesarean section fed with mother milk during were the reference group for all infants born by cesarean section.
  The breastfeeding infants were the reference group
  Interventions: Other: Breastfeeding infants
- Infants born by ED-fed fermented formula (Active Comparator): Feeding infants with fermented formula milk. Infants born by eutocic delivery were fed either with fermented formula milk or with standard formula during the first 3 months of life
  Interventions: Dietary Supplement: Feeding infants with fermented formula milk
- Infants born by ED-fed standard formula (Placebo Comparator): Feeding infants with standard formula milk. Infants born by eutocic delivery were fed either with fermented formula milk or with standard formula during the first 3 months of life
  Interventions: Other: Feeding infants with standard formula milk
- Infants born by ED-breastfed (Other): Infants born by eutocic delivery were fed either with fermented formula milk or with standard formula during the first 3 months of life.
  The breastfeeding infants were the reference group.
  Interventions: Other: Breastfeeding infants

INTERVENTIONS:
Dietary Supplement: Feeding infants with fermented formula milk — Infants enrolled were fed either with fermented formula milk or with standard formula during the first four months of life. Breastfed infants were the reference group.
  Arms: Infants born by CS-fed fermented formula; Infants born by ED-fed fermented formula
Other: Feeding infants with standard formula milk — Infants enrolled were fed either with fermented formula milk or with standard formula during the first four months of life. Breastfed infants were the reference group.
  Arms: Infants born by CS-fed standard formula; Infants born by ED-fed standard formula
Other: Breastfeeding infants — Reference group
  Arms: Infants born by CS-breastfed; Infants born by ED-breastfed

SUMMARY:
This is a single-center, double-blind, randomized controlled trial, with parallel groups and reference group. The aim of the study was to investigate whether feed a fermented formula milk leads to an increase of anti-microbial peptides such as catelecidine, alpha and beta defensins and secretory-IgA, compared to feed a standard formula (Plasmon Primigiorni), according to mode of delivery. Breastfed infants were the reference group.

DETAILED DESCRIPTION:
The microbiota plays an important role in modulating the development of the immune system, making decisive the interrelation that between nutrition, microbiota and immune cells to modulate long-term health outcomes.

The type of feeding, especially breastfeeding, and the type of delivery are factors that can contribute to the development of the microbiota. Specifically, the exclusive breastfeeding promotes the development of bifidobacteria that promotes protection against potential infections and the development of the immune system.

In recent years it was improved the biological effects of formula milk, that represent the substitutes of breast milk when this is not available or if there are contraindications to breastfeeding. Functional foods derived from fermentation of cow's milk with probiotic strains have been proposed for the prevention of infectious diseases of the child. Recently, in a monocentric double-blind prospective study, the efficacy of fermented cow's milk with Lactobacillus paracasei CBA L74 was evaluated in the prevention of common winter infections in children aged between 12 and 48 months. In this study, children treated with fermented milk had a lower incidence of respiratory and gastrointestinal tract infections compared to the control group. This effect was associated with a significant stimulation of innate immunity (α- and β-defensin, LL-37) and acquired (secretory IgA) and to a modulation of composition and function of the intestinal microbiota characterized by a significant increase in strains producing butyric acid (Firmicutes phyla). The nutritional intervention was very well accepted by the children and no adverse events were observed.

Primary objectives of this study were:

To evaluate whether the feeding with a fermented formulated milk determines an increase in anti-microbial peptides such as catelecidine, alpha and beta defensin and secretory IgA compared to the feed with the standard formula (Plasmon Primigiorni), with reference to the mother's milk.

Secondary objective:

* Value the tolerance in the two groups of infants fed with the two formulas in the study, with reference to the group of infants fed with breast milk.
* Value the modifications of the intestinal microbiota in the two groups of infants fed with the two formulas in the study, with reference to the group of infants fed with breast milk.

Study design: Single-center, randomized, double-blind, parallel group study with reference group.

Methods:

* Evaluation of the anthropometric parameters (weight, length and cranial circumference)
* Evaluation of body composition by plethysmography
* Evaluation of the gastrointestinal tolerance of fermented formulated milk by means of data collection and diary delivery to the parents of the participants
* Evaluation of the safety of fermented formulated milk by recording adverse events
* Determination of faecal samples of antimicrobial peptides (defensins, catelecidines), IgA, microbiota and metabolome.

Infants will be enrolled at birth (within 7 days of life) upon acquisition of the informed consent of both parents.

At the time of enrollment, newborns who take breast milk due to the absence of breast milk will be randomized to receive up to the third month of age or a fermented formulated milk or a standard formula (Plasmon First Days).

Enrollment will be carried out by promoting and supporting breastfeeding and, in the event of exclusive breastfeeding forecasts for at least the first 3 months of age, newborns will be included in the study as a control group.

There are 3 medical visits to enrollment (V0), the first (V1) and the third month of life (V2).

During the visits the anthropometric parameters, the body composition, and the gastroenteric tolerance will be evaluated. A stool sample will also be collected at the three points of the life study in order to determine the anti-microbial peptides (catelecidine, alpha and beta defensin) and the secretory IgA, and perform the analysis of the microbiota and the metabolome.

Statistical analysis:

The sample size was determined to identify between the two groups of infants, the one that received the fermented formulated milk and the one that received standard formulated milk (Plasmon Primigiorni), a difference in the content of faecal α-defensins on samples of feces. Considering the results of the effect of a treatment with milk fermented with L. paracasei CBA L74 on fecal α-defensins in children attending preschool centers mean value (DS) vs placebo [4.8 (4.2) vs 1 (0.6), respectively] we calculated that 12 newborns are needed per group with a power of 84% and an alpha of 0.05. Assuming a 30% drop-out rate, at least 16 newborns per group must be recruited.

Criteria for the evaluation of variables The descriptive analyzes will be performed by calculating mean, median and standard deviations for the continuous variables and expressing the distribution of the frequencies for the discrete variables. The main analysis will resort to tests for independent samples, Student or Mann-Whitney tests according to the distribution of the outcome variables. To jointly analyze the trend in time from V0 to V2 of the outcome variables in the two groups, the one that received the fermented formulated milk and the one that received the standard formula, based on the type of delivery (spontaneous or cesarean) will be used regression models for repeated measurements (random effects models or GEE models).

ELIGIBILITY:
Inclusion Criteria:

* Full term healthy infants
* Gestational age from 37 to 41 weeks
* Weight appropriate for gestational age (from 10th to 90th centile according to World Health Organization chart)
* Human milk not available or not possible

Exclusion criteria:

* Weight small for gestational age (< 10th centile) or large for gestational age (> 90th centile) according to World Health Organization chart
* Congenital abnormalities, chromosomal, hearth, gastrointestinal, respiratory, neurological or metabolic disease.
* Perinatal infections
* Positive familiarity for milk proteins allergies

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline Innate immunity at 30 days of life and at 90 days of life. | 0-7 days of life, at 30 days of life and at 90 days of life.
  Fecal dosage of catelecidines, alfa and beta defensins and sIgA

SECONDARY OUTCOMES:
Gastrointestinal tolerance | 0-7 days of life, at 30 days of life and at 90 days of life.
  Gastrointestinal tolerance was evaluated by the use of a daily diary computed by the parents to record vomiting/gaseous colics/stool frequency.
Weight | 0-7 days of life, at 30 days of life and at 90 days of life.
  weight (g)
Body composition | 0-7 days of life and at 90 days of life.
  Body composition assessment in term of fat mass and fat free mass by air displacement
Anthropometry | 0-7 days of life, at 30 days of life and at 90 days of life.
  length and head circumference (cm)
Microbiota | 0-7 days of life and at 90 days of life.
  gut microbiota assessment
Metabolomics | 0-7 days of life and at 90 days of life.
  stool metabolomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Mosca, Prof, Principal Investigator — NICU. Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Milano, Milan, Italy, 20122
Locations (1):
- Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not shared with other researchers.

REFERENCES:
- [Result] Nocerino R, Paparo L, Terrin G, Pezzella V, Amoroso A, Cosenza L, Cecere G, De Marco G, Micillo M, Albano F, Nugnes R, Ferri P, Ciccarelli G, Giaccio G, Spadaro R, Maddalena Y, Berni Canani F, Berni Canani R. Cow's milk and rice fermented with Lactobacillus paracasei CBA L74 prevent infectious diseases in children: A randomized controlled trial. Clin Nutr. 2017 Feb;36(1):118-125. doi: 10.1016/j.clnu.2015.12.004. Epub 2015 Dec 17. PMID 26732025
- [Result] Zagato E, Mileti E, Massimiliano L, Fasano F, Budelli A, Penna G, Rescigno M. Lactobacillus paracasei CBA L74 metabolic products and fermented milk for infant formula have anti-inflammatory activity on dendritic cells in vitro and protective effects against colitis and an enteric pathogen in vivo. PLoS One. 2014 Feb 10;9(2):e87615. doi: 10.1371/journal.pone.0087615. eCollection 2014. PMID 24520333
- [Result] Thibault H, Aubert-Jacquin C, Goulet O. Effects of long-term consumption of a fermented infant formula (with Bifidobacterium breve c50 and Streptococcus thermophilus 065) on acute diarrhea in healthy infants. J Pediatr Gastroenterol Nutr. 2004 Aug;39(2):147-52. doi: 10.1097/00005176-200408000-00004. PMID 15269618
- [Result] Indrio F, Ladisa G, Mautone A, Montagna O. Effect of a fermented formula on thymus size and stool pH in healthy term infants. Pediatr Res. 2007 Jul;62(1):98-100. doi: 10.1203/pdr.0b013e31806772d3. PMID 17515847
- [Derived] Roggero P, Liotto N, Pozzi C, Braga D, Troisi J, Menis C, Gianni ML, Berni Canani R, Paparo L, Nocerino R, Budelli A, Mosca F, Rescigno M. Analysis of immune, microbiota and metabolome maturation in infants in a clinical trial of Lactobacillus paracasei CBA L74-fermented formula. Nat Commun. 2020 Jun 1;11(1):2703. doi: 10.1038/s41467-020-16582-1. PMID 32483147